CLINICAL TRIAL: NCT01061359
Title: Application Of Epirubicin Within A Neo-/Adjuvant Chemotherapy In Patients With Primary Breast Cancer ((ANWENDUNGSBEOBACHTUNG,MOI 99056 -Neo-/Adjuvante Chemotherapie Des Primären Mammakarzinoms Der Frau Mit Farmorubicin®))
Brief Title: Application Of Epirubicin Within A Neo-/Adjuvant Chemotherapy In Patients With Primary Breast Cancer
Status: Completed | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer, Inc.
Other Study IDs: 378-ONC-0030-0144; A6051029/MOI99056
Record Dates: First submitted 2010-02-01; First posted 2010-02-03 (Estimated); Results first posted 2010-11-18 (Estimated); Last update posted 2010-12-29 (Estimated); Status verified 2010-12

CONDITIONS: Breast Neoplasm
Keywords: Breast Cancer; Neoadjuvant Treatment; Chemotherapy; Adjuvant; Epirubicin
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Non-Interventional Study: Chemotherapy containing Epirubicin
  Interventions: Drug: Epirubicin: Observational Study

INTERVENTIONS:
Drug: Epirubicin: Observational Study — Observational: Chemotherapy

SUMMARY:
Evaluation of efficacy of treatment with epirubicin (5 years follow-up). Evaluation of frequency of dose reduction. Evaluation of frequency of neoadjuvant treatment with E(120mg) / C(600mg). Evaluation of unexpected and serious adverse events.

(E=Epirubicin; C =Cyclophosphamide)

DETAILED DESCRIPTION:
Postmarketing surveillance study. Non-Probability Sample

ELIGIBILITY:
Inclusion Criteria:

* Pre- and postmenopausal female patients with histologically confirmed primary breast cancer

Exclusion Criteria:

* Metastatic breast cancer, locally advanced or recurrent breast cancer, previous cancer history

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Female patients with primary breast cancer
Sampling Method: Non-Probability Sample
Enrollment: 1981 (Actual)
Dates: Start 1999-01; Primary Completion 2009-10 (Actual); Study Completion 2009-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=378-ONC-0030-0144&StudyName=Application%20Of%20Epirubicin%20Within%20A%20Neo-/Adjuvant%20Chemotherapy%20In%20Patients%20With%20Primary%20Breast%20Cancer

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 1982 participants were enrolled, however, during database lock, 10 participants were identified as duplicates. Therefore, a total of 1972 unique participants were identified for the study.
Groups:
- Entire Study Population: Includes all groups enrolled in the study
Period: Overall Study
Arm/Group | Entire Study Population
Started | 1972
Completed | 670 (Completed 5 years of follow-up: 668 Disease free and 2 Relapsed)
Not Completed | 1302
Not completed — Death | 32
Not completed — Lost to Follow-up | 1072
Not completed — Relapse | 187
Not completed — Secondary neoplasm | 11

BASELINE CHARACTERISTICS:
Arm/Group | Entire Study Population
Number analyzed (Participants) | 1972
Age Continuous [Median (Full Range); unit: years] | 54.73 [25.36 to 80.42]
Age, Customized [Number; unit: participants]
  >=20 and <30 years | 12
  >=30 and <40 years | 167
  >=40 and <50 years | 512
  >=50 and <60 years | 568
  >=60 and <70 years | 557
  >=70 and <80 years | 101
  >=80 and <90 years | 1
  Unknown | 54
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1972
  Male | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Disease Free Survival (DFS)
Description: Percentage of participants with DFS who completed 5 year follow-up visit.
Time Frame: 3m, 6m, 9m, 1y, 1.5y, 2y, 2.5y, 3y, 3.5y, 4y, 4.5y, 5y
Population: Intent to treat (ITT)
Measure: Number; unit: Percentage of participants
Groups:
- Epirubicin: Includes groups enrolled to receive all treatments of epirubicin
Arm/Group | Epirubicin
Number analyzed (Participants) | 1972
Percentage of participants | 83.7

2. Secondary Outcome: Time to Progression (TTP)
Time Frame: 3m, 6m, 9m, 1y, 1.5y, 2y, 2.5y, 3y, 3.5y, 4y, 4.5y, 5y
Population: 16.3% of patients had experienced disease progression by the end of the study. As this is less than 50% the median time to progression is not defined.
Measure: Median (Full Range); unit: months
Arm/Group | Epirubicin
Number analyzed (Participants) | 0

3. Secondary Outcome: Time to Recurrence (DFI)
Time Frame: 3m, 6m, 9m, 1y, 1.5y, 2y, 2.5y, 3y, 3.5y, 4y, 4.5y, 5y
Population: Median time to recurrence was not reached.
Measure: Median (Full Range); unit: months
Arm/Group | Epirubicin
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Description: Only spontaneous adverse events were collected as reported by health care professionals. All events are reported under serious adverse events.
Arm/Group | Epirubicin
Serious Adverse Events (participants affected / at risk) | 16/1972
Other Adverse Events (participants affected / at risk) | 0/1972
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Epirubicin (N=1972)
Aneaemia (Blood and lymphatic system disorders) | 3 (3)
Leukopenia (Blood and lymphatic system disorders) | 6 (6)
Neutropenia (Blood and lymphatic system disorders) | 3 (3)
Pancytopenia (Blood and lymphatic system disorders) | 4 (4)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1)
Cardiac failure acute (Cardiac disorders) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1)
Intestinal infarction (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 2 (2)
Stomatitis (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 2 (2)
Death (General disorders) | 1 (1)
Disease progression (General disorders) | 2 (3)
General physical health deterioration (General disorders) | 1 (1)
Mucosal inflammation (General disorders) | 3 (3)
Pyrexia (General disorders) | 1 (1)
Candidiasis (Infections and infestations) | 1 (1)
Cellulitis (Infections and infestations) | 1 (1)
Mastitis (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 1 (2)
Sepsis (Infections and infestations) | 1 (1)
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (4)
Bronchial carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Metastases to nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Metastasis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2)
Ovarian cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Cerebral haemorrhage (Nervous system disorders) | 1 (1)
Nervous system disorder (Nervous system disorders) | 1 (1)
Transient ischaemic attack (Nervous system disorders) | 1 (1)
Confusional state (Psychiatric disorders) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Blister (Skin and subcutaneous tissue disorders) | 1 (1)
Thrombosis (Vascular disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.